CLINICAL TRIAL: NCT00271011
Title: A Phase II Study of Mitomycin C, Irinotecan and Cetuximab in Patients With Previously Treated, Metastatic Colorectal Cancer
Brief Title: A Study of Mitomycin C, Irinotecan, and Cetuximab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued due to the death of a co-investigator and a second co-investigator leaving the institution.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2005-060; HUM 00000749 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2005-12-27; First posted 2005-12-29 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Mitomycin; Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mitomycin C, Irinotecan and Cetuximab (Experimental): Patients will receive mitomycin C 7 mg/m2 as a bolus infusion on day -1 of each 28 day cycle.
  Patients will receive cetuximab 400 mg/m2 loading dose over 90 minutes cycle 1, day 1. All subsequent weekly cetuximab treatments will be 250 mg/m2 as a 60 minute infusion days 1, 8, 15, and 22 of each 28 day cycle.
  Patients will receive irinotecan 140 mg/m2 as a 90 minute infusion on days 1 and 15 of each 28 day cycle after cetuximab infusion. Patients found to be homozygous for UGT1A1*28 allele will receive irinotecan 110 mg/m2.
  Interventions: Drug: Mitomycin C; Drug: Cetuximab; Drug: Irinotecan.

INTERVENTIONS:
Drug: Mitomycin C — Patients will receive mitomycin C 7 mg/m2 as a bolus infusion on day -1 of each 28 day cycle.
  Other Names: Mutamycin® (trade name)
Drug: Cetuximab — Patients will receive cetuximab 400 mg/m2 loading dose over 90 minutes cycle 1, day 1. All subsequent weekly cetuximab treatments will be 250 mg/m2 as a 60 minute infusion days 1, 8, 15, and 22 of each 28 day cycle.
  Other Names: Erbitux (trade name)
Drug: Irinotecan. — Patients will receive irinotecan 140 mg/m2 as a 90 minute infusion on days 1 and 15 of each 28 day cycle after cetuximab infusion. Patients found to be homozygous for UGT1A1*28 allele will receive irinotecan 110 mg/m2.
  Other Names: Camptosar (trade name)

SUMMARY:
Colorectal cancer (CRC) is one of the more common cancers in the United States with over 145,000 new cases expected in 2005. Surgery is the main treatment for CRC. However for some who relapse after surgery, or are unable to have surgery, chemotherapy is the primary treatment for this more advanced CRC. Some chemotherapy drugs are given to the patient by themselves, but many are given in combination with other chemotherapy treatment drugs and they seem to work better together than by themselves. This study will investigate the effectiveness of the combination of three chemotherapy drugs in patients who have been previously treated for their CRC and it has returned. This study will also evaluate any rash that is associated with the drug Cetuximab. The three therapy drugs are Mitomycin C, Irinotecan, and Cetuximab.

DETAILED DESCRIPTION:
We propose a phase II trial which combines mitomycin C, irinotecan and cetuximab in patients with previously treated metastatic colorectal cancer with wild type non mutated K-Ras. The goals of this investigation are to develop an effective systemic therapy for previously treated patients with CRC with wild type K-Ras, to further explore the relationship of mitomycin C induced topoisomerase 1 gene expression and response to irinotecan, and to define and characterize the biology of cetuximab induced skin rash.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis of colorectal cancer.
2. Clinical and/or radiologic evidence of metastatic disease.
3. One previous systemic treatment for metastatic disease.
4. Age > 18.
5. Presence of at least one measurable lesion.
6. Adequate hematopoetic (absolute neutrophil count > 1500/mm3, platelet count > 100,000/mm3), renal (serum creatinine < 1.5 mg/dl), and hepatic function (bilirubin < 1.5 and transaminases < 5.0 x upper normal limit).
7. ECOG performance status 0-2.
8. Life expectancy > 3 months.
9. Patients must be informed of the investigational nature of this study and provide written informed consent in accordance with the institutional and federal guidelines prior to the initiation of therapy.

Exclusion Criteria:

1. No recognized brain metastasis.
2. No previous treatment with mitomycin C or cetuximab.
3. No other systemic malignancy requiring treatment within the past one year.
4. Pregnant or lactating women may not participate. Women/men of reproductive potential must agree to use an effective contraceptive method.
5. Patients must have no other serious medical or psychiatric illness that would limit the ability of the patient to receive protocol therapy or provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-12; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mitomycin C, Irinotecan and Cetuximab
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mitomycin C, Irinotecan and Cetuximab
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 56 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an Objective Response
Description: The primary objective of this single-arm phase II study is to determine the response rate (Percentage patients with Complete Response (CR) + Percentage of patients with Partial Response (PR)) for the combination of mitomycin C, irinotecan, and cetuximab in metastatic colorectal cancer with wild type K-Ras. Complete response will be defined as the disappearance of all measurable and evaluable disease for at least 4 weeks without the appearance of new lesions. Partial response will be defined as a decrease in the sum of the longest diameter of target lesions by at least 30% for at least 4 weeks without the appearance of any new lesions.
Time Frame: 2 months
Population: The study was discontinued and not completed due to the death of a co-investigator and a second co-investigator leaving the institution.
Arm/Group | Mitomycin C, Irinotecan and Cetuximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Patients Experiencing Hematologic and Non-hematologic Adverse Events
Description: The proportion of patients experiencing hematological and non-hematological toxicities will be summarized.
Time Frame: 2 months
Population: The study was discontinued and not completed due to the death of a co-investigator and a second co-investigator leaving the institution. Since accrual was not completed the proportion of patients experiencing toxicities could not be statistically determined.
Arm/Group | Mitomycin C, Irinotecan and Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Mitomycin C, Irinotecan and Cetuximab
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitomycin C, Irinotecan and Cetuximab (N=13)
Death, Cause Unknown (General disorders) | 1 (1)
Gastrointestinal Obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitomycin C, Irinotecan and Cetuximab (N=13)
Hemolysis (Blood and lymphatic system disorders) | 3 (3)
Fatigue (General disorders) | 9 (13)
Insomnia (Psychiatric disorders) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10 (14)
Anorexia (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (5)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Watery eye (Eye disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
The study was discontinued and not completed due to the death of a co-investigator and a second co-investigator leaving the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No